CLINICAL TRIAL: NCT03640715
Title: Validation of a Screening Tool for Social and Health Vulnerability in Pediatric Clinical Practice Tool Child Vulnerable -ENVU
Brief Title: Validation of a Screening Tool for Social and Health Vulnerability in Pediatric Clinical Practice
Acronym: ENVU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2017-28
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Infant Conditions

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A (Other): Group A: no vulnerability according to expert with no indication of any PASS marker care
  Interventions: Other: ENVU
- group B (Other): Group B: probable vulnerability according to the expert with indication of at least one PASS marker care
  Interventions: Other: ENVU
- group c (Other): Group C: high vulnerability according to the expert with indication of at least two care markers PASS
  Interventions: Other: ENVU

INTERVENTIONS:
Other: ENVU — "ENfant VUlnerable": a clinical tool for screening for social and health vulnerability in pediatrics - tool: VUlnerable Child (ENVU) -; to allow for an appropriate orientation of the patient care pathway. The metrological validation of diagnostic performances (sensitivity, specificity, positive and negative likelihood ratios) will be studied in confrontation with the opinion of an expert caregiver in the care of vulnerable populations.

SUMMARY:
In 2014, the french hospital emphasized the need for tools to screen for social fragility in order to make explicit the choices of orientation of patients. To date, caregivers do not have any tools or clinical benchmarks for individual assessment of pediatric social and health vulnerability.

The use of the Health Care Access Permanence Services (PASS) is intended to facilitate access to the health care system for people in precarious situations with care and social support within and outside the institutions. health.

The hypothesis tested is that the use of a formalized tool makes it possible to improve the detection of pediatric social vulnerability and to overcome reluctance to practice by a simple, rapid and justified approach with regard to ongoing care.

The primary objective is to validate a clinical tool for screening for pediatric social and health vulnerability - Tool: VUlnerable Child (ENVU) -; to allow for an appropriate orientation of the patient care pathway. The metrological validation of diagnostic performances (sensitivity, specificity, positive and negative likelihood ratios) will be studied in confrontation with the opinion of an expert caregiver in the care of vulnerable populations.

This multicenter cross-sectional validation study of the screening tool will be conducted in two SAUPs with a pediatric PASS.

1000 children will be included in the centers for a period of 1 year.

Following the introduction of the ENVU tool and after an expert interview, three groups of patients will be identified:

Group A: no vulnerability according to expert with no indication of any PASS marker care Group B: probable vulnerability according to the expert with indication of at least one PASS marker care Group C: high vulnerability according to the expert with indication of at least two care markers PASS Group B and C patients will be reviewed at 6 months for a second visit to the ENVU tool.

The main evaluation criterion will be the concordance between the indication of the use of the PASS by the "expert" PASS nurse (indicator of a significant social and health vulnerability) and the result of the ENVU tool.

DETAILED DESCRIPTION:
In 2014, the french hospital emphasized the need for tools to screen for social fragility in order to make explicit the choices of orientation of patients. To date, caregivers do not have any tools or clinical benchmarks for individual assessment of pediatric social and health vulnerability.

The use of the Health Care Access Permanence Services (PASS) is intended to facilitate access to the health care system for people in precarious situations with care and social support within and outside the institutions. health.

The hypothesis tested is that the use of a formalized tool makes it possible to improve the detection of pediatric social vulnerability and to overcome reluctance to practice by a simple, rapid and justified approach with regard to ongoing care.

The primary objective is to validate a clinical tool for screening for pediatric social and health vulnerability - Tool: VUlnerable Child (ENVU) -; to allow for an appropriate orientation of the patient care pathway. The metrological validation of diagnostic performances (sensitivity, specificity, positive and negative likelihood ratios) will be studied in confrontation with the opinion of an expert caregiver in the care of vulnerable populations.

The secondary objectives will be to study the validity of the ENVU tool with regard to pathologies epidemiologically associated with social vulnerability: hypotrophy, prematurity, weight-loss disorders, school delay, asthma, skin infection, oral health, visual disturbances not treatment, delayed immunization, over-consumption of unscheduled care in SAUP, iron deficiency and lead poisoning (if research indicated by the reason for consultation). The illustration of the added value of the PASS care will be observed by a before-after study of the ENVU tool and the collected clinical data.

This multicenter cross-sectional validation study of the screening tool will be conducted in two SAUPs with a pediatric PASS.

1000 children will be included in the centers for a period of 1 year.

Following the introduction of the ENVU tool and after an expert interview, three groups of patients will be identified:

Group A: no vulnerability according to expert with no indication of any PASS marker care Group B: probable vulnerability according to the expert with indication of at least one PASS marker care Group C: high vulnerability according to the expert with indication of at least two care markers PASS Group B and C patients will be reviewed at 6 months for a second visit to the ENVU tool.

The main evaluation criterion will be the concordance between the indication of the use of the PASS by the "expert" PASS nurse (indicator of a significant social and health vulnerability) and the result of the ENVU tool.

ELIGIBILITY:
Inclusion Criteria:

* from 3 to 15 years old,
* And consultant in the SAUP and PASS services investigators,
* And outside periods of custody and affluence,
* And accompanied by at least one parent or guardian
* And accepting to participate.

Exclusion Criteria:

* Consultation in SAUP during the period of guard or affluence,
* Or Patient who has already consulted at PASS,
* Or child who has already participated in the study,
* Or in the absence of any parent (father or mother),
* Or current child protection measure - or evoked by doctors during the stay at SAUP,
* Or parents who do not speak French and can not translate at the moment of inclusion,
* Or inclusion of another child of the siblings,
* Or refusal of the child or parents,
* Or impossibility to organize an interview with an expert caregiver during the stay at the SAUP without prolonging it.

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1000 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Number of patient for whom expertise is in good accordance with ENVU tool | 1 days
  The main evaluation criterion will be the concordance between the indication of the use of the PASS by the caretaker of the "expert" PASS (indicator of a significant social and health vulnerability) and the result of the ENVU tool.

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France

REFERENCES:
- [Derived] Laporte R, Babe P, Jouve E, Daguzan A, Mazoue F, Minodier P, Noel G, Urbina D, Gentile S. Developing and Validating an Individual-Level Deprivation Index for Children's Health in France. Int J Environ Res Public Health. 2022 Dec 16;19(24):16949. doi: 10.3390/ijerph192416949. PMID 36554830